CLINICAL TRIAL: NCT03978182
Title: Accelerated Deep TMS in the Elderly Depressed: A Brain Imaging Approach
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: replaced by other study
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-190
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2019-06

CONDITIONS: Old Age; Depression
Keywords: repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: geriatric depressed patients after randomization at time T1 (on a Monday for MRI) will be divided into two groups to receive 20 sessions of real or sham adTMS treatment respectively. A given patient who first received active treatment will not receive sham, because of the carry-over effects; a patient who first received sham treatment now receives active adTMS in an open phase. This treatment will be spread over the four succeeding afternoons (5 daily sessions). In the second week, strictly the same treatment schedule will be followed but with the reverse order. A second brain imaging assessment will be performed exactly 1 week after the first week (time T2) and a third time scan exactly after 2 weeks (time T3).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: unblinding will be done after the first week, in this way subjects receiving sham will have the opportunity to receive active treatment in the second week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active accelerated deep rTMS (Active Comparator): Stimulation: We will use a Magstim Rapid2 Plus1 Magnetic Stimulator connected to a Brainsway H1 coil, which includes a sham option. In analogy to our former accelerated rTMS studies (2, 3), all patients will receive 20 dTMS sessions (5 sessions per day; 4 consecutive days) with a stimulation intensity of 120% of the subject's resting MT, as reported by Levkovitz et al.(4). Furthermore, we selected these FDA approved dTMS parameters, so that for one session each dTMS repetition includes 2-sec pulse trains separated by 20-sec inter-train intervals. Patients will receive 55 trains in each treatment session, for a total of 1980 pulses per session. This makes 9900 pulses/day, and in total 39600 pulses per treatment.
  Interventions: Device: accelerated deep rTMS
- sham (Sham Comparator): Built-in sham in the H1 Helmet (same device as active treatment)
  Interventions: Device: accelerated deep rTMS

INTERVENTIONS:
Device: accelerated deep rTMS — A Magstim Rapid2 Plus1 Magnetic Stimulator connected to the Brainsway dTMS system with the H1-coil investigational device (Brainsway Ltd, Jerusalem, Israel). The coil is situated inside a helmet to achieve effective cooling during stimulation. A sham coil is also included in the same helmet. The sham coil mimics scalp sensations and the acoustic artifact of the active stimulation without inducing neuronal activation.

SUMMARY:
With a growing number of elderly persons, geriatric depression - associated with important morbidity and mortality- is becoming a significant health problem. Given the risk of polypharmacy and increased side effects, alternative non pharmaceutical treatments such as repetitive transcranial magnetic stimulation (rTMS) may be a solution. Given recent positive results with accelerated rTMS in the elderly depressed, it is of interrest to continue to develop promising non-invasive treatment stimulations. The FDA approved deep brain TMS (dTMS) technique may be a promising option, targeting the brain underneath the neocortex with potentially better response and remission rates. Therefore, in a sham-controlled cross-over fashion, the investigators will treat 44 geriatric depressed patients with accelerated dTMS (5 sessions/day over 4 days only), and evaluate clinical efficacy and safety. Because new introduced rTMS paradigms should be rigorously neurobiologically examined before applying them on a regular basis, this research will include multimodal brain imaging techniques to elucidate the working mechanisms of this application in order to optimize treatment for such populations.

DETAILED DESCRIPTION:
An initially double-blind sham-controlled cross-over study in geriatric depressed patients to investigate whether accelerated (a)dTMS is a safe and effective clinical option for this cohort. After the first week evaluations and MRI, there will be an open label phase in which patients who did receive active treatment in the first week will not receive any further rTMS sessions, those patients who had received sham however will get their active treatment in the second week. The independent researcher will use the treatment allocation list to inform the investigators if an active treatment faze is needed in the second week.

ELIGIBILITY:
Inclusion Criteria:

* In and outpatients (age 65 year or older) meeting Diagnostic and Statistical Manual of Mental Disorders (DSM 5) criteria for unipolar depression according 17-item Hamilton depression rating scale (HDRS-17) score of 17 or more, who failed to respond to at least one adequate course with an antidepressant medication trial, including the current one. Stable current antidepressant treatment (>6 weeks) will be continued during the stimulation.
* Able to read, understand and sign the Informed Consent Form.

Exclusion Criteria:

* Psychosis (exception: depression with psychotic features)
* A personal history of seizures or epilepsy, a history of seizures or epilepsy in first degree relatives and the presence of any known factor that can lower the seizure threshold (sleep deprivation, abuse substance, etc.), previous head injury and the presence of metallic implants in the cephalic region (e.g., aneurysm clips, shunts, stimulators, cochlear implants, electrodes) with the exception of dental fillings and the presence of cardiac pacemakers, neurostimulators, surgical clips or other electronic equipment, comorbidity with some neurological disorders: increased intracranial pressure, space-occupying lesion, history of stroke or transient ischemic attack, brain aneurysm.
* Patients with cognitive disturbances or dementia will not be included (Mini Mental State) < 24.
* Suicide attempt within 6 months before the start of the study or present risk of Suicide with the Columbia-Suicide Severity Rating Scale (C-SSRS).
* ECT exposure (current major depressive episode)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | During 1 week (and 2 weeks for patients who received sham in the first week)
  Number of participants with treatment-related adverse events as assessed by questionning the patient on each stimulation day
clinical efficacy measured by change in the 17 item Hamilton Depression rating Scale score. | from screening until last visit (week 4)
  for a total score between 0 and 48, the higher the total score the more severe the depression. Used measures are : for response (reduction from baseline of ≥ 50% in the total score) and remission (total HAMD-17 score ≤ 7)
clinical efficacy measured by change in the Beck-Inventory of Depression-II score | from screening until last visit (week 4)
  for a total score between 0 and 63, the higher the total score the more severe the depression. A score of ≤9 is the criterion for remission, and BDI-II score decrease of 50% from baseline is the criterion for treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Baeken, MD Phd, Study Director — Universitair Ziekenhuis Brussel

IPD SHARING:
Plan to Share IPD: No